CLINICAL TRIAL: NCT02596581
Title: Association of Gingival Crevicular Fluid Chemerin and IL-6 Levels in Chronic Periodontitis With and Without Type 2 Diabetes Mellitus After Non-Surgical Periodontal Therapy
Brief Title: Chemerin and IL-6 Levels in Diabetes and Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Asisstant Proffessor, Bulent Ecevit University, Bulent Ecevit University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-116-17-06
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus
Keywords: periodontitis; diabetes mellitus; chemerin; interleukin-6
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- diabetics with periodontally healthy group (No Intervention): Control group
- systemically and periodontally healthy group (No Intervention): Control group
- diabetics with chronic periodontitis group (Active Comparator): non-surgical periodontal treatment was performed
  Interventions: Other: non-surgical periodontal treatment
- chronic periodontitis group (Active Comparator): non-surgical periodontal treatment was performed
  Interventions: Other: non-surgical periodontal treatment

INTERVENTIONS:
Other: non-surgical periodontal treatment — scaling and root planing were performed
  Arms: chronic periodontitis group; diabetics with chronic periodontitis group

SUMMARY:
The aims of the present study were to determine the gingival crevicular fluid (GCF) chemerin and interleukin-6 (IL-6) levels and to analyse the relationship between chemerin and IL-6 in periodontal health and in chronic periodontitis (CP) with and without type 2 diabetes mellitus (T2DM) as well as to evaluate the effect of non-surgical periodontal therapy on the GCF chemerin levels.

DETAILED DESCRIPTION:
Adipose tissue is an active endocrine organ that secretes several inflammatory cytokines, namely, adipokines, which interfere with insulin sensitivity, with glucose and lipid metabolism, and with the inflammatory process.Chemerin, a more recently identified adipose tissue specific adipokine, has a crucial role in adipocyte differentiation and development, as well as in glucose, lipid metabolism and inflammation. Experimental data supports both pro- and anti-inflammatory roles for chemerin in immune cells. Therefore, it is not clear whether chemerin contributes more to the progression of inflammation or the resolution.The present investigation has been devoted to elucidate the role of chemerin in the pathogenesis that might link between DM and periodontal disease. We hypothesize that chemerin may hold value as an inflammatory mediator in CP patients with and without T2DM and non-surgical periodontal treatment could have a beneficial influence on the levels of chemerin.

The aim of this study were:

1. to determine the role of chemerin in the pathogenesis of periodontal disease and DM via comparing with GCF levels of IL-6, which has a known proinflammatory effect in periodontal disease and DM
2. to evaluate the effect of non-surgical periodontal treatment on GCF chemerin levels in periodontitis patients with and without T2DM.

The study included eighty subjects: 20 subjects with systemically and periodontally healthy (CTRL group), 20 patients with T2DM and periodontally healthy (DM-CTRL group), 20 patients with systemically healthy and CP (CP group), 20 patients with CP and T2DM (DM-CP group). Periodontitis patients received nonsurgical periodontal therapy. GCF sampling and clinical periodontal parameters were assessed at baseline and 6 weeks after periodontal therapy. Chemerin and interleukin-6 (IL-6) levels were measured by enzyme-linked immunosorbent assay, and their relative ratios were calculated.

Subjects were clinically evaluated using the following parameters; plaque index (PI), gingival index (GI) , PD, clinical attachment level (CAL) and BOP (deemed positive if it occurred within 15 seconds after probing). Clinical measurements were recorded by one calibrated examiner at six sites per tooth from the full-mouth teeth excluding third molars using with a Williams periodontal probe (Nordent Manufacturing Inc., ElkGrove Village, IL, USA) calibrated in millimeters. Anthropometric measurements included weight (kg) and height (m) of the subjects to calculate the BMI ( weight divided by the square of height, kg/m2 ).

All clinical and radiological examinations, sampling site selections were performed by one examiner and the samples were collected on the day after clinical examination of patients. This was to prevent contamination of GCF with blood associated with the probing of inflamed sites. The deepest two pocket sites of single-rooted teeth were selected for the collection of GCF in both periodontitis groups, and also two pocket sites with an absence of inflammation were sampled to ensure the collection of an adequate amount of GCF in control groups. In patients from CP and DM-CP groups, sites showing greatest PD when measured with a periodontal probes and signs of inflammation, along with radiographic conformation of bone loss were sampled. GCF samples were collected at baseline and after 8 weeks from baseline sampling in both periodontitis groups, and only at baseline in control groups. To avoid salivary contamination, the sites to be sampled were rinsed with water, isolated by cotton rolls and gently air dried. Paper strips (Periopaper; Oraflow Inc.,Smithtown, NY, USA) were gently inserted 1-2 mm into the sulcus/pocket for 30 seconds. Care was taken to avoid mechanical injury of the gingival tissues. All samples containing blood and saliva were discarded. The two strips from two sites of each individual were placed into coded sealed plastic eppendorf tubes and pooled before freezing at -80 degree

ELIGIBILITY:
Inclusion Criteria:

* Diabetic subjects should have T2DM and had no any known systemic diseases other than T2DM
* Subjects who had HbA1c levels < 8% and ≥ 6.5% (well and moderate control)
* Chronic periodontitis patients had radiographic evidence of bone loss and attachment loss with a minimum of 6 teeth having pocket probing depth (PD) ≥ 5mm in at least 2 different quadrants
* Control groups were designed as healthy if the full-mouth probing depth (PD) was ≤3mm and bleeding on probing (BOP) score < %15 at examination and they had no radiographic evidence of alveolar bone loss.

Exclusion Criteria:

* Presence of other systemic disorders that could influence the course of periodontal disease; pregnancy, lactation, current and former use of tobacco;
* Administration of non-steroidal and anti-inflammatory drugs or antibiotic therapies within the previous 6 months;
* Need for antibiotic prophylaxis for dental treatment and having received non-surgical periodontal treatment within the past 6 months or surgical periodontal treatment within the past 12 months.
* Subjects who had body mass index (BMI) >24.9 kg /m2

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
gingival crevicular fluid chemerin level | 8th weeks
  gingival crevicular fluid chemerin levels change from baseline to at 8th weeks

SECONDARY OUTCOMES:
Interleukin-6 | 8th weeks
  change of gingival crevicular fluid IL-6 levels from baseline at 8th weeks
gingival index | 8ths week
  gingiva inflammation score
plaque index | 8ths week
  oral hygiene score
bleeding on probing | 8th weeks
  deemed positive if it occurred within 15 seconds after probing
clinical attachment level | 8th weeks
  distance between the cemento-enamel junction to the deepest point of periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Umut Ballı, Phd, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Figen Öngöz Dede, Phd, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Şeyma Bozkurt Doğan, Phd, DDS, Study Chair — Bülent Ecevit University Faculty of Dentistry; Erdim Sertoğlu, MD, DDS, Principal Investigator — Elazig Military Hospital, Department of Medical Biochemistry, Elazığ, Turke